CLINICAL TRIAL: NCT03887312
Title: Development, Piloting and Evaluation of a Phone-Delivered Psychological Intervention (t-CETA) for Syrian Refugee Children in Lebanon: Phase II
Brief Title: Phone-Delivered Psychological Intervention (t-CETA) for Mental Health Problems in 8-17 Year-Old Syrian Refugee Children
Acronym: t-CETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Médecins du Monde (Other); American University of Beirut Medical Center (Other); Johns Hopkins University (Other); Medical School Hamburg (Other)
Responsible Party: Principal Investigator, Michael Pluess, Professor of Developmental Psychology, Head of Psychology Department, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ReDA_012540; 28371 (Other Grant/Funding Number: ELRHA)
Record Dates: First submitted 2019-01-25; First posted 2019-03-22 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Depression; Anxiety; PTSD; Conduct Disorder; Oppositional Defiant Disorder
Keywords: Phone-delivered therapy; Cognitive behavioral therapy (CBT); Telephone-delivered therapy; Children; Adolescents; Syrian refugees
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Conduct Disorder; Oppositional Defiant Disorder

STUDY DESIGN:
Intervention Model Description: There are two arms in the RCT, t-CETA and treatment as usual (TaU), to which children will be randomly assigned. A stratified randomization model will be used, with randomization occurring within four separate groups:
  1. Males aged 8-12 years
  2. Males aged 13-17 years
  3. Females aged 8-12 years
  4. Females aged 13-17 years
  A third group will consist of participants who do not wish to be randomised, but who will receive t-CETA. Their data will not form part of the RCT but will be used to provide additional data on efficacy, implementation, and acceptability of t-CETA.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will not be blind to treatment allocation. The team providing treatment and conducting in-session assessments will not be blind to treatment allocation.
  One individual will be responsible for processing raw data and hence will not be blind as to treatment allocation.
  The team carrying out independent assessments will be blind to treatment allocation.
  The investigator team carrying out data analysis will be blind to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- t-CETA (Experimental): Telephone-delivered Common Elements Treatment Approach (t-CETA). t-CETA sessions of up to 30 minutes will be delivered 1-2 times per week for approximately 8-12 weeks. The number and content of sessions will be tailored to each child, thus there will be some variation.
  Interventions: Behavioral: t-CETA
- Médecins du Monde treatment as usual (Active Comparator): Treatment as usual provided by Médecins du Monde. The number and content of sessions will vary depending on the needs of the child.
  Interventions: Behavioral: Médecins du Monde treatment as usual

INTERVENTIONS:
Behavioral: t-CETA — Cognitive Behavioural Therapy (CBT) based approach delivered over the telephone. Components are available for common problems, including anxiety, depression, PTSD, conduct problems, substance abuse, and safety issues (including self-harm or suicidal ideation), and a tailored treatment package is produced for each child based on the presenting problem(s) and response to treatment. There are components for use with both child and caregiver.
  Other Names: Telephone-delivered Common Elements Treatment Approach
  Arms: t-CETA
Behavioral: Médecins du Monde treatment as usual — Case manager-led care, with referral to a psychotherapist or psychiatrist as necessary. Médecins du Monde's approach is based on a joint collaboration between mental health trained case managers (who undergo extensive training by experts in the field on topics including Psychological First Aid, Child Protection, Gender Based Violence, etc.) and psychotherapists from different schools (providing Eye Movement Desensitization and Reprocessing [EMDR] for trauma, Interpersonal Therapy [IPT] for depression, Cognitive Behavioural Therapy [CBT], motivational counselling, familial or systemic therapy, and integrative approaches). Thus the number and content of sessions, and the person delivering treatment (case manager, psychotherapist, psychiatrist) vary.
  Arms: Médecins du Monde treatment as usual

SUMMARY:
This study evaluates the effectiveness of t-CETA, a version of Common Elements Treatment Approach (CETA) adapted to be delivered over the telephone, in treating common mental health problems in 8-17 year old Syrian refugee children living in Lebanon. Children will be randomly assigned to receive either t-CETA or treatment as usual provided by Médecins du Monde, an NGO providing medical and mental health services to Syrian refugees in Lebanon. If families do not agree to randomisation, they will be offered t-CETA and their data will be used to evaluate implementation and acceptability of the intervention.

Symptoms of common mental health problems, including anxiety, depression, PTSD, and behavioural problems, and psychological well-being, will be measured before treatment, immediately after treatment, and three months after treatment is completed. Groups will be compared to determine if t-CETA is at least as effective as standard treatment provided by Médecins du Monde.

DETAILED DESCRIPTION:
Common Elements Treatment Approach (CETA) is a transdiagnostic treatment approach designed to treat common mental health problems such as anxiety, depression, post-traumatic stress disorder (PTSD), and externalising behaviour problems. It uses a Cognitive Behavioural Therapy (CBT) approach and has been used in both adults and children. There are a number of different components that can be put together to provide a treatment approach that is tailored to each individual. For this study CETA has been adapted to be delivered over the telephone (t-CETA).

The overall study has two specific objectives:

1. Development of telephone-delivered CETA (t-CETA) by adapting the scientifically validated face-to face CETA programme (including manual and detailed training material). This was completed during Phase I.
2. Scientific evaluation of the effectiveness of t-CETA applying a randomized controlled clinical trial. This will be completed during Phase II and is described in the remainder of this submission.

Study design:

The implementation and efficacy of t-CETA will be tested with a randomized controlled clinical trial. Up to 120 Syrian refugee children will be randomly allocated to either t-CETA or treatment as usual provided by Médecins du Monde in primary healthcare centres in the Beqaa valley. Clinical interviews with children and primary caregivers will be conducted before the intervention to determine suitability for inclusion. Assessments will be carried out before and after the intervention as well as during a 3-month follow-up assessment by independent trained enumerators blind to study condition. If families do not agree to randomisation, they will be offered t-CETA only and their data will be used to carry out additional evaluation of efficacy, implementation and acceptability of the intervention. Implementation and acceptance of the intervention will be further assessed with a qualitative study based on interviews with a subset of involved Syrian refugee children, their caregivers as well as mental health staff.

Sample:

Children included in the study will be selected from the large sample of an NICHD funded study on the biological pathways of risk and resilience in Syrian refugee children based in Lebanon headed by PI Prof. Michael Pluess and co-PI Prof. Elie Karam ("Biological Pathways of Risk and Resilience in Syrian Refugee Children" [BIOPATH]; Sponsor: Queen Mary University of London [ReDA Ref: 011120]; Ethical approval: Institutional Review Board of the University of Balamand, Lebanon [Ref: IRB/O/024-16/1815] and Ministry of Public Health in Lebanon, in consultation with the Lebanese National Consultative Committee on Ethics). BIOPATH is a longitudinal study and includes 1,600 Syrian refugee families in the Beqaa valley. For each of these children there is data on a range of psychological outcomes (PTSD, depression, anxiety, externalising behavioural problems). From the 1,600 children, the investigators will select up to 120 based on psychological symptoms assessed routinely as part of the BIOPATH study. If insufficient numbers of children from the BIOPATH study are recruited, the following additional approaches will be used: (i) children from BIOPATH who take part in the linked VaST study (which involves completing the MINI KID clinical interview) will be approached if they meet inclusion criteria and are interested in accessing mental health services; (ii) other children in the families who took part in BIOPATH (e.g., siblings and cousins) and for whom families requested mental health services will be approached; (iii) referrals will be accepted from other agencies; (iv) information sessions will be conducted in the community (e.g., in Informal Tented Settlements) to inform families about the research and allow them to request mental health assessment for their child(ren); (v) families in contact with participating families will be able to contact the study for information and to request mental health assessment for their child (snowballing approach).

Recruitment:

Primary caregivers will be contacted over the phone and offered clinical assessment for their child at no cost, as part of routine clinical care. Families will be invited to attend an appointment at an MdM clinic or be visited at home for this assessment. Families who attend the appointment will first undertake a brief interview to establish the presenting problem. Following this and providing children do not meet exclusion criteria, they will be offered inclusion in the t-CETA study. Those who do not want to participate in research, or who clearly meet exclusion criteria, will be offered a standard clinical intake assessment and treatment as usual provided by Médecins du Monde. Those who do want to participate in research will complete the informed consent process, and a clinical interview (Mini-International Neuropsychiatric Interview For Children And Adolescents; MINI KID) and severity score (Clinical Global Impression severity score; CGI-s) will then be used to guide whether children meet inclusion criteria. Those who do not meet inclusion criteria or whose difficulties are not appropriate for CETA will be offered treatment as usual by Médecins du Monde or referral to another agency, as appropriate.

Following recruitment, participants will complete the first in-session assessment (see below for assessment details) and be prepared for baseline assessments. A visual aids booklet will be provided to assist with responding to questionnaire items and the child and caregiver will have the opportunity to answer practice questions using the visual aids.

The baseline independent assessment will then be conducted via phone (see below for assessment details).

Randomization and blinding:

Following baseline independent assessment participants will be randomized to either t-CETA or treatment as usual (TaU) provided by Médecins du Monde (MdM). Stratified randomization will be used by randomizing within each of the following four groups:

1. Males aged 8-12 years
2. Males aged 13-17 years
3. Females aged 8-12 years
4. Females aged 13-17 years

Participants and the treatment teams will not be blind to treatment allocation. The team carrying out independent assessments and the team carrying out data analysis will be blind to treatment allocation.

If participants do not agree to randomisation, they will be offered t-CETA only; treatment and data collection will be identical to that described for children receiving t-CETA as part of the RCT.

Treatment:

t-CETA: Children will receive telephone delivered therapy 1 or 2 times per week for up to 30 minutes per session. Treatment will take approximately 8-16 weeks. There will be some variation in the number and content of treatment sessions because t-CETA will be tailored to each participant depending on the presenting problem(s).

TaU: Children will receive case manager-led care, involving initial assessment by a case manager, with intervention then provided by a case manager, and/or referral to a psychotherapist or psychiatrist as necessary. Médecins du Monde's approach is based on a joint collaboration between mental health trained case managers (who undergo extensive training by experts in the field on topics including Psychological First Aid, Child Protection, Gender Based Violence, etc.) and psychotherapists from different schools (providing Eye Movement Desensitization and Reprocessing [EMDR] for trauma, Interpersonal Therapy [IPT] for depression, Cognitive Behavioural Therapy [CBT], motivational counselling, familial or systemic therapy, and integrative approaches). Thus the number and content of sessions, and the person delivering treatment (case manager, psychotherapist, psychiatrist) will vary.

Supervision:

Both t-CETA and TaU teams will be closely supervised by experienced clinical psychologists. Supervision will occur during weekly sessions, with more frequent supervision for challenging cases and to manage safety issues.

Independent Assessments:

Trained assessors will be independent of the treatment team and blind to treatment condition. They will conduct assessments over the phone (or face-to-face if phone assessment is not possible). This will take approximately 30-45 minutes per child and 30-45 minutes per caregiver. The assessment includes standardized questionnaires about the child's symptoms and adaptive functioning. Participants will have the option to use the visual aids booklet provided to help them respond to questions. Data will be entered into the online platform Qualtrics, uploaded to a secure server. Participants will only be identified using an ID on Qualtrics; identifying details will not be entered. The assessment process will be supervised by a qualified clinical psychologist (Local PI, Dr Tania Bosqui).

Independent assessments will be conducted at baseline (pre-treatment), immediately following treatment, and at three months follow-up.

In-session assessment:

The case managers providing treatment will conduct these assessments, hence they will not be blind to treatment condition.

Client Monitoring Form (CMF): The CMF is a key part of t-CETA treatment: it is intended to guide selection of t-CETA components and monitor progress. It is a questionnaire measure and is developed to be specific to each population in which CETA or t-CETA is used. In this study it will also be used with children receiving TaU. It will be administered at baseline and then weekly at the beginning of treatment sessions.

PSYCHLOPS: This questionnaire will be used during the first treatment session, during the session that is the approximate mid-point, and the final session.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-17 years, male or female
2. Live with a parent or other legal guardian
3. Child and/or parent identifies that the child has mental health difficulties and requests services
4. At high risk of having a mental disorder as indexed by falling in the top 40% of the distribution in any one of the following child-report questionnaires: (i) Screen for Child Anxiety Related Emotional Disorders (SCARED), (ii) Center for Epidemiological Studies Depression Scale for Children (CES-DC), (iii) Child PTSD Symptom Scale (CPSS); AND falling in the top 40% of the distribution in the following parent report questionnaire: Strengths and Difficulties Questionnaire (SDQ) total difficulties [Criterion 4 is only applicable to children for whom these data are available from participation in the BIOPATH study; Criterion 5 takes precedence over Criterion 4 where both are available]
5. Confirmation of significant level of symptoms and functional impairment on clinical interview (MINI KID) as indicated by (i) meeting full or probable diagnostic criteria for ANY of the following: any category of mood disorder, any category of anxiety disorder, PTSD, conduct disorder, or oppositional defiant disorder; AND (ii) Clinical Global Impression severity (CGI-s) score of >3
6. Parent/legal guardian gives informed consent and child gives assent to take part

Exclusion Criteria:

1. Problem for which t-CETA would not be appropriate, including psychiatric disorders for which CETA treatment is not recommended (e.g., bipolar disorder, psychosis), severe distress (e.g., acute suicidal ideation), or problems that would preclude delivery over the telephone (e.g., selective mutism)
2. Parent or legal guardian is not able to provide consent
3. Child protection issues (e.g., acute maltreatment) that are judged by clinician to make trial inclusion inappropriate
4. Any inclusion criteria not met

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Emotional and behavioural problem composite score | Baseline (pre-treatment)
  Measures common emotional and behavioural problems in children. Scores from the following questionnaire measures will be aggregated: Child PTSD Symptom Scale (CPSS; child self-report), Center for Epidemiological Studies Depression Scale for Children (CES-DC; child self-report), Screen for Child Anxiety Related Emotional Disorders (SCARED; child self-report), the Strengths and Difficulties Questionnaire (SDQ; parent report) externalising score, and conduct disorder / oppositional defiant disorder items (caregiver report). Arabic versions of all questionnaires are used. Scores on these questionnaires have been divided into deciles based on data from the population from which the study sample is drawn and each decile is converted into a score ranging from 0 (lowest decile) to 9 (highest decile). These decile scores are then summed for the four questionnaire measures, giving a total score ranging from 0 to 36. Higher scores indicate greater problems.
Emotional and behavioural problem composite score | Approximately 12 weeks (immediately after treatment has been completed)
  Measures common emotional and behavioural problems in children. Scores from the following questionnaire measures will be aggregated: Child PTSD Symptom Scale (CPSS; child self-report), Center for Epidemiological Studies Depression Scale for Children (CES-DC; child self-report), Screen for Child Anxiety Related Emotional Disorders (SCARED; child self-report), the Strengths and Difficulties Questionnaire (SDQ; parent report) externalising score, and conduct disorder / oppositional defiant disorder items (caregiver report). Arabic versions of all questionnaires are used. Scores on these questionnaires have been divided into deciles based on data from the population from which the study sample is drawn and each decile is converted into a score ranging from 0 (lowest decile) to 9 (highest decile). These decile scores are then summed for the four questionnaire measures, giving a total score ranging from 0 to 36. Higher scores indicate greater problems.
Emotional and behavioural problem composite score | Approximately 24 weeks (3 months following completion of treatment)
  Measures common emotional and behavioural problems in children. Scores from the following questionnaire measures will be aggregated: Child PTSD Symptom Scale (CPSS; child self-report), Center for Epidemiological Studies Depression Scale for Children (CES-DC; child self-report), Screen for Child Anxiety Related Emotional Disorders (SCARED; child self-report), the Strengths and Difficulties Questionnaire (SDQ; parent report) externalising score, and conduct disorder / oppositional defiant disorder items (caregiver report). Arabic versions of all questionnaires are used. Scores on these questionnaires have been divided into deciles based on data from the population from which the study sample is drawn and each decile is converted into a score ranging from 0 (lowest decile) to 9 (highest decile). These decile scores are then summed for the four questionnaire measures, giving a total score ranging from 0 to 36. Higher scores indicate greater problems.
World Health Organization Disability Assessment Schedule for Children (WHODAS-Child, adapted): child report | Baseline (pre-treatment)
  WHODAS-child orginally adapted for Rwanda and then translated into Arabic for use with Syrian children (child self-report). Measures three domains of functional impairment: getting along with people, life activities (ability to carry out responsibilities at home and school), and participation in society (ability to engage in community, civil and recreational activities). Subscales are averaged to produce a Global Disability score. Scores are expressed as a percentage so range from 0-100, with higher scores indicating greater impairment.
World Health Organization Disability Assessment Schedule for Children (WHODAS-Child, adapted): child report | Approximately 12 weeks (immediately after treatment has been completed)
  WHODAS-child orginally adapted for Rwanda and then translated into Arabic for use with Syrian children (child self-report). Measures three domains of functional impairment: getting along with people, life activities (ability to carry out responsibilities at home and school), and participation in society (ability to engage in community, civil and recreational activities). Subscales are averaged to produce a Global Disability score. Scores are expressed as a percentage so range from 0-100, with higher scores indicating greater impairment.
World Health Organization Disability Assessment Schedule for Children (WHODAS-Child, adapted): child report | Approximately 24 weeks (3 months following completion of treatment)
  WHODAS-child orginally adapted for Rwanda and then translated into Arabic for use with Syrian children (child self-report). Measures three domains of functional impairment: getting along with people, life activities (ability to carry out responsibilities at home and school), and participation in society (ability to engage in community, civil and recreational activities). Subscales are averaged to produce a Global Disability score. Scores are expressed as a percentage so range from 0-100, with higher scores indicating greater impairment.
World Health Organization Disability Assessment Schedule for Children (WHODAS-Child, adapted): caregiver report | Baseline (pre-treatment)
  WHODAS-child orginally adapted for Rwanda and then translated into Arabic for use with Syrian children (caregiver report). Measures three domains of functional impairment: getting along with people, life activities (ability to carry out responsibilities at home and school), and participation in society (ability to engage in community, civil and recreational activities). Subscales are averaged to produce a Global Disability score. Scores are expressed as a percentage so range from 0-100, with higher scores indicating greater impairment.
World Health Organization Disability Assessment Schedule for Children (WHODAS-Child, adapted): caregiver report | Approximately 12 weeks (immediately after treatment has been completed)
  WHODAS-child orginally adapted for Rwanda and then translated into Arabic for use with Syrian children (caregiver report). Measures three domains of functional impairment: getting along with people, life activities (ability to carry out responsibilities at home and school), and participation in society (ability to engage in community, civil and recreational activities). Subscales are averaged to produce a Global Disability score. Scores are expressed as a percentage so range from 0-100, with higher scores indicating greater impairment.
World Health Organization Disability Assessment Schedule for Children (WHODAS-Child, adapted): caregiver report | Approximately 24 weeks (3 months following completion of treatment)
  WHODAS-child orginally adapted for Rwanda and then translated into Arabic for use with Syrian children (caregiver report). Measures three domains of functional impairment: getting along with people, life activities (ability to carry out responsibilities at home and school), and participation in society (ability to engage in community, civil and recreational activities). Subscales are averaged to produce a Global Disability score. Scores are expressed as a percentage so range from 0-100, with higher scores indicating greater impairment.

SECONDARY OUTCOMES:
Child PTSD Symptom Scale (CPSS) | Baseline (pre-treatment)
  Child PTSD Symptom Scale, Arabic version, child self-report. Total post-traumatic stress disorder symptom scores range from 0-51 and higher scores indicate a higher level of symptoms.
Child PTSD Symptom Scale (CPSS) | Approximately 12 weeks (immediately after treatment has been completed)
  Child PTSD Symptom Scale, Arabic version, child self-report. Total post-traumatic stress disorder symptom scores range from 0-51 and higher scores indicate a higher level of symptoms.
Child PTSD Symptom Scale (CPSS) | Approximately 24 weeks (3 months following completion of treatment)
  Child PTSD Symptom Scale, Arabic version, child self-report. Total post-traumatic stress disorder symptom scores range from 0-51 and higher scores indicate a higher level of symptoms.
Center for Epidemiological Studies Depression Scale for Children (CES-DC) | Baseline (pre-treatment)
  Center for Epidemiological Studies Depression Scale for Children, Arabic 10-item version, child-self-report. Total depression symptom scores range from 0-30 and higher scores indicate a higher level of symptoms.
Center for Epidemiological Studies Depression Scale for Children (CES-DC) | Approximately 12 weeks (immediately after treatment has been completed)
  Center for Epidemiological Studies Depression Scale for Children, Arabic 10-item version, child-self-report. Total depression symptom scores range from 0-30 and higher scores indicate a higher level of symptoms.
Center for Epidemiological Studies Depression Scale for Children (CES-DC) | Approximately 24 weeks (3 months following completion of treatment)
  Center for Epidemiological Studies Depression Scale for Children, Arabic 10-item version, child-self-report. Total depression symptom scores range from 0-30 and higher scores indicate a higher level of symptoms.
Screen for Child Anxiety Related Emotional Disorders (SCARED) | Baseline (pre-treatment)
  Screen for Child Anxiety Related Emotional Disorders, Arabic 18-item version, child-self-report. Total anxiety symptoms scores range from 0-36 and higher scores indicate a higher level of symptoms.
Screen for Child Anxiety Related Emotional Disorders (SCARED) | Approximately 12 weeks (immediately after treatment has been completed)
  Screen for Child Anxiety Related Emotional Disorders, Arabic 18-item version, child-self-report. Total anxiety symptoms scores range from 0-36 and higher scores indicate a higher level of symptoms.
Screen for Child Anxiety Related Emotional Disorders (SCARED) | Approximately 24 weeks (3 months following completion of treatment)
  Screen for Child Anxiety Related Emotional Disorders, Arabic 18-item version, child-self-report. Total anxiety symptoms scores range from 0-36 and higher scores indicate a higher level of symptoms.
Externalising behaviour problems score | Baseline (pre-treatment)
  Score derived from the Strengths and Difficulties Questionnaire (SDQ; parent-report) externalising score (10 items) and items measuring behaviours associated with conduct disorder (CD) and oppositional defiant disorder (ODD) (12 items). Arabic version, caregiver report. The SDQ externalising score ranges from 0-20 and the CD/ODD items range from 0-24. These will be summed to given an externalising behaviour problems score ranging from 0-44 and higher scores indicate a higher level of problems.
Externalising behaviour problems score | Approximately 12 weeks (immediately after treatment has been completed)
  Score derived from the Strengths and Difficulties Questionnaire (SDQ; parent-report) externalising score (10 items) and items measuring behaviours associated with conduct disorder (CD) and oppositional defiant disorder (ODD) (12 items). Arabic version, caregiver report. The SDQ externalising score ranges from 0-20 and the CD/ODD items range from 0-24. These will be summed to given an externalising behaviour problems score ranging from 0-44 and higher scores indicate a higher level of problems.
Externalising behaviour problems score | Approximately 24 weeks (3 months following completion of treatment)
  Score derived from the Strengths and Difficulties Questionnaire (SDQ; parent-report) externalising score (10 items) and items measuring behaviours associated with conduct disorder (CD) and oppositional defiant disorder (ODD) (12 items). Arabic version, caregiver report. The SDQ externalising score ranges from 0-20 and the CD/ODD items range from 0-24. These will be summed to given an externalising behaviour problems score ranging from 0-44 and higher scores indicate a higher level of problems.
WHO-5 Well-Being Index (WHO-5) | Baseline (pre-treatment)
  WHO-5 Well-Being Index, Arabic version, child-self-report. Total well-being scores range from 0-100 and higher scores indicate higher well-being.
WHO-5 Well-Being Index (WHO-5) | Approximately 12 weeks (immediately after treatment has been completed)
  WHO-5 Well-Being Index, Arabic version, child-self-report. Total well-being scores range from 0-100 and higher scores indicate higher well-being.
WHO-5 Well-Being Index (WHO-5) | Approximately 24 weeks (3 months following completion of treatment)
  WHO-5 Well-Being Index, Arabic version, child-self-report. Total well-being scores range from 0-100 and higher scores indicate higher well-being.
Youth Life Orientation Test (YLOT) | Baseline (pre-treatment)
  Youth Life Orientation Test, measuring optimism, Arabic 4-item version, child self-report.
  Total optimism scores range from 0-12 and higher scores indicate higher optimism.
Youth Life Orientation Test (YLOT) | Approximately 12 weeks (immediately after treatment has been completed)
  Youth Life Orientation Test, measuring optimism, Arabic 4-item version, child self-report.
  Total optimism scores range from 0-12 and higher scores indicate higher optimism.
Youth Life Orientation Test (YLOT) | Approximately 24 weeks (3 months following completion of treatment)
  Youth Life Orientation Test, measuring optimism, Arabic 4-item version, child self-report.
  Total optimism scores range from 0-12 and higher scores indicate higher optimism.
PSYCHLOPS Pre-Therapy (Kids or Teen) | At first treatment session, approximately 1-2 weeks after baseline
  Psychological Outcome Profiles (PSYCHLOPS) Pre-Therapy, Kids version (for children aged 8-12 years), Teen version (for age 13-16 years). Arabic version, child self-report. Three subscale scores are used, Problems (range 0-4 [Kids], 0-10 [Teen]), Functioning (range 0-4 [Kids], 0-5 [Teen]), and Wellbeing (range 0-4 [Kids], 0-5 [Teen]). These are summed to give a total score (range 0-12 [Kids], 0-20 [Teen]). Scores from the Kids version will be scaled to be equivalent to the Teen version so scores are comparable across both age groups. Higher scores indicate greater problems, impaired functioning, and poorer wellbeing.
PSYCHLOPS During Therapy (Kids or Teen) | At mid-point treatment session, approximately 5-6 weeks after baseline
  Psychological Outcome Profiles (PSYCHLOPS) During Therapy, Kids version (for children aged 8-12 years), Teen version (for age 13-16 years). Arabic version, child self-report. Three subscale scores are used, Problems (range 0-4 [Kids], 0-10 [Teen]), Functioning (range 0-4 [Kids], 0-5 [Teen]), and Wellbeing (range 0-4 [Kids], 0-5 [Teen]). These are summed to give a total score (range 0-12 [Kids], 0-20 [Teen]). Scores from the Kids version will be scaled to be equivalent to the Teen version so scores are comparable across both age groups. Higher scores indicate greater problems, impaired functioning, and poorer wellbeing.
PSYCHLOPS Post-Therapy (Kids or Teen) | At final treatment session, approximately 8-12 weeks after baseline
  Psychological Outcome Profiles (PSYCHLOPS) Post-Therapy, Kids version (for children aged 8-12 years), Teen version (for age 13-16 years). Arabic version, child self-report. Three subscale scores are used, Problems (range 0-4 [Kids], 0-10 [Teen]), Functioning (range 0-4 [Kids], 0-5 [Teen]), and Wellbeing (range 0-4 [Kids], 0-5 [Teen]). These are summed to give a total score (range 0-12 [Kids], 0-20 [Teen]). Scores from the Kids version will be scaled to be equivalent to the Teen version so scores are comparable across both age groups. Higher scores indicate greater problems, impaired functioning, and poorer wellbeing.
Client Monitoring Form (CMF) | Baseline (pre-treatment)
  Client Monitoring Form developed for this study to measure mental health problems, substance use, and safety issues during treatment, Arabic version, child self-report.
Client Monitoring Form (CMF) | Final treatment session, approximately 8-12 weeks after baseline
  Client Monitoring Form developed for this study to measure mental health problems, substance use, and safety issues during treatment, Arabic version, child self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pluess, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Medecins du Monde, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murray LK, Dorsey S, Haroz E, Lee C, Alsiary MM, Haydary A, Weiss WM, Bolton P. A Common Elements Treatment Approach for Adult Mental Health Problems in Low- and Middle-Income Countries. Cogn Behav Pract. 2014 May;21(2):111-123. doi: 10.1016/j.cbpra.2013.06.005. PMID 25620867
- [Background] Murray LK, Hall BJ, Dorsey S, Ugueto AM, Puffer ES, Sim A, Ismael A, Bass J, Akiba C, Lucid L, Harrison J, Erikson A, Bolton PA. An evaluation of a common elements treatment approach for youth in Somali refugee camps. Glob Ment Health (Camb). 2018 Apr 25;5:e16. doi: 10.1017/gmh.2018.7. eCollection 2018. PMID 29868236
- [Background] Bolton P, Lee C, Haroz EE, Murray L, Dorsey S, Robinson C, Ugueto AM, Bass J. A transdiagnostic community-based mental health treatment for comorbid disorders: development and outcomes of a randomized controlled trial among Burmese refugees in Thailand. PLoS Med. 2014 Nov 11;11(11):e1001757. doi: 10.1371/journal.pmed.1001757. eCollection 2014 Nov. PMID 25386945
- [Background] Weiss WM, Murray LK, Zangana GA, Mahmooth Z, Kaysen D, Dorsey S, Lindgren K, Gross A, Murray SM, Bass JK, Bolton P. Community-based mental health treatments for survivors of torture and militant attacks in Southern Iraq: a randomized control trial. BMC Psychiatry. 2015 Oct 14;15:249. doi: 10.1186/s12888-015-0622-7. PMID 26467303
- [Derived] Pluess M, McEwen FS, Biazoli C, Chehade N, Bosqui T, Skavenski S, Murray L, Weierstall-Pust R, Bolton P, Karam E. Delivering therapy over telephone in a humanitarian setting: a pilot randomized controlled trial of common elements treatment approach (CETA) with Syrian refugee children in Lebanon. Confl Health. 2024 Sep 20;18(1):58. doi: 10.1186/s13031-024-00616-2. PMID 39304918
- [Derived] McEwen FS, El Khatib H, Hadfield K, Pluess K, Chehade N, Bosqui T, Skavenski S, Murray L, Weierstall-Pust R, Karam E, Pluess M. Feasibility and acceptability of phone-delivered psychological therapy for refugee children and adolescents in a humanitarian setting. Confl Health. 2024 Jan 13;18(1):7. doi: 10.1186/s13031-023-00565-2. PMID 38218936

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT03887312/Prot_SAP_001.pdf